CLINICAL TRIAL: NCT02247791
Title: Study of Prosthesis Choice in Older Patients With a Dislocated Femoral Neck Fracture of the Hip
Brief Title: Uncemented Compared to Cemented Femoral Stems in Total Hip Arthroplasty
Acronym: CHANCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Danderyd Hospital (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Principal Investigator, Olof Skoldenberg, Director of research, Orthopaedic dept, Danderyd Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHANCE
Record Dates: First submitted 2013-10-21; First posted 2014-09-25 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cemented femoral stem (Active Comparator): Patient undergoing total hip arthroplasty surgery
  Interventions: Procedure: Cemented femoral stem
- Uncemented femoral stem (Active Comparator): Patients undergoing total hip arthroplasty
  Interventions: Procedure: Uncemented femoral stem

INTERVENTIONS:
Procedure: Uncemented femoral stem — All patients will be randomized to operation with either an uncemented femoral stem or a cemented femoral stem
  Other Names: BiMetric uncemented femoral stem
  Arms: Uncemented femoral stem
Procedure: Cemented femoral stem — All patients will be randomized to operation with either an uncemented femoral stem or a cemented femoral stem
  Other Names: CPT cemented femoral stem
  Arms: Cemented femoral stem

SUMMARY:
The purpose of this study is to evaluate whether an uncemented hip prosthesis is as safe as an cemented hip prosthesis for patients undergoing total hip arthroplasty surgery following a displaced femoral neck fracture.

DETAILED DESCRIPTION:
The study will randomize patients between an uncemented and cemented stem

ELIGIBILITY:
Inclusion Criteria:

* Acute Displaced femoral neck fracture
* Subject is aged between 65-79 years
* Independent walker with or without walking aides
* Subject is able and capable of providing consent to participate in the study

Exclusion Criteria:

* Patients with Rheumatoid Arthritis
* Patients with an impaired cognitive dysfunction
* Patients with Pathological fractures
* Patients with substance abuse
* Patients with fracture older than 36-hours on arrival at the A&E
* Patients suffering from cancer
* Patients determined by principal investigator to be unsuitable for inclusion

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2009-09; Primary Completion 2016-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Hip related complication rate | 2 years
  All hip-related complications
Health-related Quality of Life | 2 years
  Health related quality of life

SECONDARY OUTCOMES:
Duration of surgery | 2 years
Intraoperative bleeding | 2 years
Hip function | 2 years
  Measured with Harris hip score

CONTACTS AND LOCATIONS:
Overall Officials: Ghazi Chammout, MD, Principal Investigator — Dept of Orthopaedics, Danderyd Hospital, Stockholm, Sweden
Locations (1):
- Danderyd Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Chammout G, Muren O, Boden H, Salemyr M, Skoldenberg O. Cemented compared to uncemented femoral stems in total hip replacement for displaced femoral neck fractures in the elderly: study protocol for a single-blinded, randomized controlled trial (CHANCE-trial). BMC Musculoskelet Disord. 2016 Sep 20;17(1):398. doi: 10.1186/s12891-016-1253-y. PMID 27646142